CLINICAL TRIAL: NCT04029571
Title: Effect and Safety of Fasting-Mimicking Diet Combined With a "Dispelling Dampness" Meal Replacement in Phlegm-Dampness Type Overweight/Obesity Patients: A Randomized Controlled Study(EASTAR)
Brief Title: Effect and Safety of TCM-FMD in Phlegm-Dampness Type Overweight/Obesity Patients(EASTAR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yuanqi Zhao,MD, Clinical Professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tcmfmd
Record Dates: First submitted 2019-07-20; First posted 2019-07-23 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Obesity
Keywords: Obesity; Fasting-mimicking diet; Traditional Chinese medicine
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TCM-FMD (Experimental): Apply fastening-mimicking diet combined with a "dispelling dampness" meal replacement. For the convenience of implementation, a cycle of 4 weeks. The first 5 days of each cycle is the calorie restriction stage (daily calorie about 800kcal). The traditional Chinese medicine with dampness effect is used as the main source of calories in this stage. The normal diet is carried out under the guidance of a professional dietitian for the next 23 days. Study for 12 weeks.
  Interventions: Drug: TCM-FMD
- FMD (Active Comparator): A "grain package" is used to replace the "dispelling dampness" meal replacement, and the other thing is the same as the proposal in TCM-FMD.
  Interventions: Other: FMD
- Normal diet (No Intervention): Carrying out normal diet under the guidance of a dietitian, for 12 weeks.

INTERVENTIONS:
Drug: TCM-FMD — Apply fastening-mimicking diet combined with a "dispelling dampness" meal replacement. For the convenience of implementation, a cycle of 4 weeks. The first 5 days of each cycle is the calorie restriction stage (daily calorie about 800kcal). The traditional Chinese medicine with dampness effect is used as the main source of calories in this stage. The normal diet is carried out under the guidance of a professional dietitian for the next 23 days. Study for 12 weeks.
  Arms: TCM-FMD
Other: FMD — A "grain package" is used to replace the "dispelling dampness" meal replacement, and the other thing is the same as the proposal in TCM-FMD.
  Arms: FMD

SUMMARY:
The primary aim of this study is to is to determine if a diet (TCM-FMD) which combine fasting-mimicking diet (FMD) with "dispelling dampness" meal replacement (a meal replacement made up of traditional Chinese medicine) is the effective dietary strategy for treatment of phlegm-dampness type overweight/obese patients. A three months randomized trial will be used to observe weight loss generated by TCM-FMD and FMD. And a group keeping a normal diet will be set as a blank control. Through comparison, we aim at examining the effects of interventions on weight and metabolic disease risk factors (plasma lipids, fasting glucose, blood pressure) The secondary aim of this study is to evaluate the safety of TCM-FMD.

DETAILED DESCRIPTION:
Background:Fasting-mimiking Diet (FMD) is a plant-based diet designed to attain fasting-like effect, firstly proposed on 2015[1]. It requires people to limit calorie intake for 5 continuous days, and then return to their normal diet after completion about 25 days until the next cycle. In a clinical trial[2], three FMD cycles reduced body weight, trunk and body fat, and reduced blood pressure, fasting blood glucose, triglycerides and total cholesterol. On the other hand, in the theory of physique of TCM theory, overweight/obesity is usually considered to be phlegm-dampness type.

Objective: We assume that using medicinal-edible plants which was considered to dispel dampness(such as fuling, shanyao, etc.) as FMD's proprietary formulations can enhance the effect of FMD on improve people's characteristic features of metabolic syndrome.

Methods: A 12-week, single-center, pilot study will be conducted to test the study objectives.A new diet is carried. It is a fasting-mimicking diet combined with a "dispelling dampness" meal replacement. Because the theory of applying traditional Chinese medicine combined with FMD, we call it TCM-FMD, the main ingredient of the "wet diet" meal package is millet. Brown rice, oats, purple sweet potato, alfalfa, yam, hazelnut, etc. For comparison, we also designed FMD to make some cereals (including millet, purple potato, oatmeal, walnut, etc.) without a moisturizing effect into a "grain package" as a control group. Both groups were administered using the FMD diet model. At the same time, a group of normal diets was also designed as a blank control group. The primary outcome measure for the study was weight; secondary outcome measures included: waist circumference, blood pressure, triglycerides, total cholesterol and fasting blood glucose, quality of life (evaluated by physical fitness scale and SF-36); safety indicators included: liver and kidney Features, etc. Both groups were subjected to caloric restriction (5 days, daily calorie about 800kcal) and normal diet (dietitian for healthy diet guidance), and the blank control group was given a normal diet.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as overweight / obesity according to the "China Adult Obesity Prevention and Treatment Expert Consensus"
* Diagnosis as phlegm-dampness type according to the "Traditional Chinese Medicine Classification and Judgment" scale published by the Chinese Medicine Association
* 18 years old ≤ age ≤ 65 years old
* Signed the informed consent

Exclusion Criteria:

* Those who have special food requirements or having a history of food allergies
* Those who have history of previous diabetes, or body weight loss, BMI ≤ 18
* Those who have had cardiovascular and cerebrovascular events within half a year, or who have a major history of surgery
* Pregnant or lactating woman
* Those who have severe primary diseases such as liver or kidney diseases, as well as abnormalities in the hematopoietic system and mental disorders
* Those who need to take special drugs (such as hormones)
* Those who refuse to provide information required for research (such as personal information, blood samples, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Body weight | Change from baseline to day 6/week 4/week 12
  Measuring the fasting weight of the day at the required time point and measured by the same instrument

SECONDARY OUTCOMES:
Triglycerides | Change from baseline to week 4/week 12
  Measured by GPO-PAP enzymatic method
Fasting glucose | Change from baseline to week 4/week 12
  Measured by Hexokinase
Blood pressure | Change from baseline to week 4/week 12
  Measure by the same sphygmomanometer

CONTACTS AND LOCATIONS:
Overall Officials: Yuanqi Zhao, MD, Study Director — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China